CLINICAL TRIAL: NCT01020760
Title: Pilot Study of Prone Posturing Following Phacovitrectomy for Thickness Macular Hole
Brief Title: Protocol for RCT of Posturing in Phacovitrectomy for Full Thickness Macular Hole (FTMH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, David Yorston, Consultant Ophthalmologist, NHS Greater Glasgow and Clyde
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version 1
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Full Thickness Macular Hole
Keywords: Macular hole; Vitrectomy; Prone posturing
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No posture (No Intervention): Patients will undergo routine phacoemulsification, pars plana vitrectomy, ILM peel and gas fluid exchange with 14% C3F8. They will be advised to avoid supine posturing for seven days after surgery, but will not be advised to posture in the face down or prone position.
- Face down posture (Experimental): Patients will undergo routine phacoemulsification, pars plana vitrectomy, ILM peel and gas fluid exchange with 14% C3F8. They will be advised to posture in the face down or prone position for 50 minutes per hour for seven days.
  Interventions: Behavioral: Face down posture

INTERVENTIONS:
Behavioral: Face down posture — Patients are requested to maintain a strict face down posture for 50 minutes out of every hour for seven days after surgery.
  Arms: Face down posture

SUMMARY:
The purpose of this study is to determine the effect of postoperative posturing on the outcome of macular hole surgery. Current practice is divided; some individuals are advised to posture face-down for 10 days and others are advised that posturing is unnecessary. By evaluating the effect of posturing in a prospective randomised controlled trial the investigators hope to determine best practice, enabling surgeons and patients to make informed decisions regarding postoperative management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having surgery for idiopathic full thickness macular hole
2. Able and willing to posture face-down for 10 days postoperatively
3. Agree to participate in the trial and able to give informed consent

Exclusion Criteria:

1. History of visual loss suggesting a duration of macular hole greater than 12 months
2. Patients unable or unwilling to posture face-down for 10 days postoperatively
3. History of trauma that may have been causative
4. Age less than 16 years (in practice idiopathic macular hole is extremely rare in patients under 30 years).
5. Previous vitrectomy surgery
6. Additional retinal breaks occurring during surgery that necessitate post-operative posturing to prevent retinal detachment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
estimate variance and effect size order to inform power calculations for further studies. | one year

SECONDARY OUTCOMES:
visual acuity and complications | one year
estimate recruitment rate and establish protocol/procedure | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Gartnavel General Hospital, Glasgow, United Kingdom

REFERENCES:
- [Result] Yorston D, Siddiqui MA, Awan MA, Walker S, Bunce C, Bainbridge JW. Pilot randomised controlled trial of face-down posturing following phacovitrectomy for macular hole. Eye (Lond). 2012 Feb;26(2):267-71. doi: 10.1038/eye.2011.220. Epub 2011 Sep 23. Erratum In: Eye (Lond). 2012 Feb;26(2):341. PMID 21941363